CLINICAL TRIAL: NCT02012998
Title: An Open-label, Controlled, Multi-centre Study of the Immunogenicity and Safety of a Challenge Dose of HBVAXPRO to Explore the Anamnestic Immune Response in Healthy Children Vaccinated 10 Years Ago With a Primary Series (3 Doses) of Either HEXAVAC or INFANRIX HEXA
Brief Title: Study of the Immunogenicity and Safety of a Challenge Dose of HBVAXPRO in Healthy Children Vaccinated 10 Years Ago With 3 Doses of HEXAVAC or INFANRIX HEXA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HXV02C; 2013-001602-28 (EudraCT Number)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Virus Diseases; Hepatitis B
MeSH Terms: conditions — Virus Diseases; Hepatitis B | interventions — Hepatitis B Vaccines; DNA, Ribosomal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HBVAXPRO Challenge dose (Experimental): HBVAXPRO 5µg
  Interventions: Biological: HBVAXPRO 5µg

INTERVENTIONS:
Biological: HBVAXPRO 5µg — 0.5mL intramuscular injection
  Other Names: Hepatitis B vaccine (rDNA)

SUMMARY:
To evaluate the immune response to Hepatitis B virus in children who have been primed with HEXAVAC or INFANRIX HEXA 10 years ago.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child
* Child vaccinated with 3 doses of HEXAVAC or 3 doses of INFANRIX HEXA as infant
* Child vaccinated with the third dose of HEXAVAC or INFANRIX HEXA at least 10 years prior to challenge dose

Exclusion Criteria:

* Receipt of more than 3 doses of any Hepatitis B containing vaccine
* History of clinical diagnosis of infection due to Hepatitis B
* History or current close contact with known carriers of Hepatitis B virus
* Prior known sensitivity or allergy to any component of HBVAXPRO
* Chronic illness / medical condition that could interfere with study conduct or completion
* Coagulation disorder that would contraindicate intramuscular injection
* Subject is pregnant
* Receipt of corticosteroids for more than 14 days in the 30 days prior to study
* Receipt of Immunoglobulins, blood or blood-derived products in the 3 months prior to study
* Planned participation in another clinical study

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 751 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with an anti-hepatitis B concentration ≥10 mIU/mL | One month after the challenge dose

SECONDARY OUTCOMES:
Percentage of subjects with an anti-hepatitis B concentration ≥10 mIU/mL | Prior to challenge dose (At Day 0 prior to administration of the challenge dose)
Solicited injection-site adverse reactions and pyrexia | Day 0 to day 4 after vaccination
Unsolicited injection-site adverse reactions and systemic adverse events | Day 0 to day 14 after vaccination
Serious adverse events | From signature of the informed consent to the last visit of the subject, an expected average of one month

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (10):
- Italy (10):
  - Sanofi Pasteur MSD Investigational Site 004, Bologna
  - Sanofi Pasteur MSD Investigational Site 009, Cagliari
  - Sanofi Pasteur MSD Investigational Site 005, Capannori
  - Sanofi Pasteur MSD Investigational Site 003, Chiavari
  - Sanofi Pasteur MSD Investigational Site 002, Latisana
  - Sanofi Pasteur MSD Investigational Site 008, Massafra
  - Sanofi Pasteur MSD Investigational Site 006, Nocera Inferiore
  - Sanofi Pasteur MSD Investigational Site 010, Ragusa
  - Sanofi Pasteur MSD Investigational Site 007, Salerno
  - Sanofi Pasteur MSD Investigational Site 001, Sassari

REFERENCES:
- [Derived] Zanetti A, Desole MG, Romano L, d'Alessandro A, Conversano M, Ferrera G, Panico MG, Tomasi A, Zoppi G, Zuliani M, Thomas S, Soubeyrand B, Eymin C, Lockhart S. Safety and immune response to a challenge dose of hepatitis B vaccine in healthy children primed 10years earlier with hexavalent vaccines in a 3, 5, 11-month schedule: An open-label, controlled, multicentre trial in Italy. Vaccine. 2017 Jul 13;35(32):4034-4040. doi: 10.1016/j.vaccine.2017.05.047. Epub 2017 Jun 16. PMID 28624307